CLINICAL TRIAL: NCT02765412
Title: Implementing Guidelines for Shared Decision Making in Lung Cancer Screening (QUE 15-286)
Brief Title: PrOVE QUERI Project #1
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: QUX 16-003; QUE 15-286 (Other Grant/Funding Number: HSR&D QUERI)
Record Dates: First submitted 2016-05-05; First posted 2016-05-06 (Estimated); Results first posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Prevention and Control
Keywords: decision support; patient preferences; risk adjustment
MeSH Terms: conditions — Patient Preference

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- standard implementation: Webinar, Promotion, Tool Access, academic detailing + Audit and Feedback
  Interventions: Other: Webinar, Promotion, and Tool Access; Other: Audit and Feedback; Other: Academic Detailing
- intensive implementation: Webinar, Promotion, and Tool Access, academic detailing + Audit and Feedback + LEAP
  Interventions: Other: Webinar, Promotion, and Tool Access; Other: LEAP; Other: Audit and Feedback; Other: Academic Detailing

INTERVENTIONS:
Other: Webinar, Promotion, and Tool Access — All sites will receive a professionally developed, 15-minute webinar that describes the tool's development (e.g., how the algorithm was designed) and a tutorial on how to use the web-site. The investigators will promote the webinar and using the tool through key local leaders. A web-link to use the tool will be placed within the lung cancer screening clinical reminder.
Other: LEAP — Sites randomized to intensive implementation will be offered participation in the LEAP program. LEAP (Learn. Engage. Act. Program) is a multi-week, online learning collaborative using systems redesign techniques to help sites identify and overcome barriers to implementation of shared decision making (use of the Decision Precision tool).
  Groups: intensive implementation
Other: Audit and Feedback — Providers at all sites will have access to this system. It will provide feedback on the screening and shared decision making process (e.g., number of provider's eligible patients screened for lung cancer, use of the tool, patient knowledge and satisfaction from patient surveys).
  Other Names: A&F
Other: Academic Detailing — All sites will be offered an academic detailing approach to implementation of Lung Decision Precision. A trained detailer will travel to all sites who agree to a visit. The detailer will meet with individual primary care providers whenever possible, and groups of providers as necessary. He will present evidence for a risk-based approach to screening and how to use the tool with patients to make tailored screening recommendations.
  Other Names: AD

SUMMARY:
The overall goal of this project is to test two strategies for implementing a shared decision making tool to be used by providers while talking to patients about lung cancer screening. Eight participating sites will be randomized to compare standard implementation with intensive implementation. Additionally, the investigators will determine the factors that were most important for successful implementation of the shared decision making tool. Finally, the investigators will survey patients to evaluate the effects of Decision Precision on patient's knowledge of the risks and benefits of lung cancer screening, the quality of their decision making, and their satisfaction with care.

DETAILED DESCRIPTION:
The overall goal of this quality improvement project is to test two strategies for implementing shared decision making, which incorporates the Decision Precision lung cancer screening tool. The investigators will use multi-site, cluster-based randomization to compare standard implementation with intensive implementation. Additionally, the investigators will determine the factors that were most important for successful implementation of the shared decision making tool. Finally, the investigators will have a human subjects research component to evaluate the effects of Decision Precision on patient's knowledge of the risks and benefits of lung cancer screening, the quality of their decision making, and their satisfaction with care.

ELIGIBILITY:
Inclusion Criteria:

* Patients at participating sites without documented exclusions for lung cancer screening who have had initial lung cancer screening clinical reminders resolved during the recruitment period

Exclusion Criteria:

Exclusions for initial lung cancer screening clinical reminders:

* history of lung, pancreatic, liver or esophageal cancer
* a health factor on file indicating they have a life expectancy of less than 6 months or who already had a chest CT in the past 12 months

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients at participating sites, age 55 to 80 years, who have a 30 pack-year smoking history and currently smoke or have quit within the past 15 years.
Sampling Method: Non-Probability Sample
Enrollment: 17033 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanner Caverly, MD MPH, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (8):
- United States (8):
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lowery J, Fagerlin A, Larkin AR, Wiener RS, Skurla SE, Caverly TJ. Implementation of a Web-Based Tool for Shared Decision-making in Lung Cancer Screening: Mixed Methods Quality Improvement Evaluation. JMIR Hum Factors. 2022 Apr 1;9(2):e32399. doi: 10.2196/32399. PMID 35363144

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eight VA sites participated in this Quality Improvement Project. Four were randomized to each arm. The number of participants in each arm reflects how many Veterans at the sites randomized to each arm who were eligible for lung cancer screening according to CDW data between October 2016 and December 2019.
Groups:
- Standard Implementation: Promotion, Tool Access, academic detailing + Audit and Feedback
  Promotion, and Tool Access: All sites will be given access to a You Tube video that describes the tool's development (e.g., how the algorithm was designed) and a tutorial on how to use the web-site. The investigators will promote the webinar and using the tool through key local leaders. A web-link to use the tool will be placed within the lung cancer screening clinical reminder.
  Audit and Feedback: Sites will be provided with reports to provide feedback on the screening and shared decision making process. Site teams were encouraged to send these reports to providers.
  Academic Detailing: All sites will be offered an academic detailing approach to implementation of Lung Decision Precision. A trained detailer will travel to all sites who agree to a visit. The detailer will meet with individual primary care providers whenever possible, and groups of providers as necessary. He will present evidence for a risk-based approach to screening and how to use the tool with patients to make tailored screening recommendations.
- Intensive Implementation: Promotion, and Tool Access, academic detailing + Audit and Feedback + LEAP
  Promotion, and Tool Access: All sites will be given access to a You Tube video that describes the tool's development (e.g., how the algorithm was designed) and a tutorial on how to use the web-site. The investigators will promote the webinar and using the tool through key local leaders. A web-link to use the tool will be placed within the lung cancer screening clinical reminder.
  LEAP: Sites randomized to intensive implementation will be offered participation in the LEAP program. LEAP (Learn. Engage. Act. Program) is a multi-week, online learning collaborative using systems redesign techniques to help sites identify and overcome barriers to implementation of shared decision making (use of the Decision Precision tool).
  Audit and Feedback: Sites will be provided with reports to provide feedback on the screening and shared decision making process. Site teams were encouraged to send these reports to providers.
  Academic Detailing: All sites will be offered an academic detailing approach to implementation of Lung Decision Precision. A trained detailer will travel to all sites who agree to a visit. The detailer will meet with individual primary care providers whenever possible, and groups of providers as necessary. He will present evidence for a risk-based approach to screening and how to use the tool with patients to make tailored screening recommendations.
Period: Overall Study
Arm/Group | Standard Implementation | Intensive Implementation
Started | 5275 | 11758
Completed | 4793 | 10903
Not Completed | 482 | 855
Not completed — Death | 482 | 855

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Implementation | Intensive Implementation | Total
Number analyzed (Participants) | 5275 | 11758 | 17033
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2373 | 6303 | 8676
  >=65 years | 2902 | 5455 | 8357
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [60 to 70] | 64 [57 to 69] | 64 [58 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196 | 848 | 1044
  Male | 5079 | 10910 | 15989
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 59 | 165 | 224
  Not Hispanic or Latino | 4904 | 10951 | 15855
  Unknown or Not Reported | 312 | 642 | 954
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 60 | 112 | 172
  Asian | 5 | 27 | 32
  Native Hawaiian or Other Pacific Islander | 27 | 63 | 90
  Black or African American | 314 | 1903 | 2217
  White | 4369 | 8788 | 13157
  More than one race | 28 | 58 | 86
  Unknown or Not Reported | 472 | 807 | 1279
Travel Distance [Median (Inter-Quartile Range); unit: miles] — Distance from Veteran's home to the VAMC where their Pack Year Clinical Reminder was completed (based on longitude and latitude).
  miles | 37.8 [13.0 to 90.2] | 45.9 [13.4 to 91.4] | 43.8 [13.3 to 91.2]

OUTCOME MEASURES:

1. Primary Outcome: Odds Ratio of the Interaction Between Lung Cancer Risk and Implementation Arm
Description: First, we estimated screening's net benefit for an individual based on their baseline lung cancer risk, as estimated using the Bach et. al. annual lung cancer incidence model. Patients are considered "high benefit" if their annual lung cancer risk is between 0.3%-1.3%. Patients outside this range are considered "preference sensitive". We fit a multilevel logistic regression model where receipt of screening is the outcome. Precision decision making is reflected in the association between baseline lung cancer risk and screening utilization: an increase in screening utilization for those at higher lung cancer risk indicates some degree of precision decision making. The primary outcome for the cluster-randomized design assesses the difference in precision decision making in the standard vs. intensive implementation arms. This is estimated as the effect on screening receipt of the interaction between risk and implementation arm.
Time Frame: post implementation, an average of 15 months
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Standard Implementation | Intensive Implementation
Number analyzed (Participants) | 5275 | 11758
odds ratio | 1.03 [0.89 to 1.19] | 1.53 [1.41 to 1.61]
Statistical Analysis 1: Comparison: Standard Implementation vs Intensive Implementation; Test type: Other — multilevel model; p = 0.081, Regression, Logistic — Two-sided test; the a priori threshold being 0.05; Adjusts for age, gender, race, comorbidities, implementation group, travel distance, and VAMC indicator; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.58 to 0.78] — OR corresponding to the interaction between implementation group and lung cancer risk, a ratio of odds ratios. The OR for screening based on lung cancer risk in the SI group versus the OR for screening based on lung cancer risk in the II group

2. Primary Outcome: Patient Satisfaction With Decision and Process
Description: Obtained from patient surveys (for the subset of the overall participants who returned surveys). The unit of measurement is one unit on the scale [scale of 0 (very poor) to 10 (very good)].
Time Frame: Survey mailed to Veteran several weeks after identified as having an initial discussion about lung cancer screening using VA administrative data
Population: Surveys were sent to eligible Veterans, the overall number of participants analyzed is a reflection of the subset of the overall participants who returned surveys. The unit of measurement is one unit on the scale [scale of 0 (very poor) to 10 (very good)].
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard Implementation | Intensive Implementation
Number analyzed (Participants) | 649 | 1451
units on a scale | 7 [3 to 9] | 7 [4 to 10]
Statistical Analysis 1: Comparison: Standard Implementation vs Intensive Implementation; Simple t-test comparing mean satisfaction ratings between arms; Test type: Other; p = 0.35, t-test, 2 sided — Two-sided test; the a priori threshold being 0.05; Median Difference (Net) = -0.15, 95% CI 2-sided [-0.16 to 0.46] — Satisfaction rating on a scale of 0 to 10; Difference is Arm 1 - Arm 2

3. Secondary Outcome: Number of Tool Assessments Where Patient Decision Aid Was Printed
Description: Number of times during study duration where patient decision aid was printed from the Lung Decision Precision web-site.
Time Frame: post implementation, up to 25 months
Population: Unable to complete - para data from website did not collect this information as planned.
Arm/Group | Standard Implementation | Intensive Implementation
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Times Dynamic Pictograph Depicting Personalized Benefit and Harm Was Opened for Display
Description: Number of times dynamic pictograph depicting personalized benefit and harm was opened for display in the Lung Decision Precision web-site during the study period, collected as para data from Decision Precision web-site
Time Frame: post implementation, up to 25 months
Population: The para data from the website is not reliable - unable to assess this planned outcome.
Groups:
- Standard Implementation: Webinar, Promotion, Tool Access, academic detailing + Audit and Feedback
  Webinar, Promotion, and Tool Access: All sites will receive a professionally developed, 15-minute webinar that describes the tool's development (e.g., how the algorithm was designed) and a tutorial on how to use the web-site. The investigators will promote the webinar and using the tool through key local leaders. A web-link to use the tool will be placed within the lung cancer screening clinical reminder.
  Audit and Feedback: Providers at all sites will have access to this system. It will provide feedback on the screening and shared decision making process (e.g., number of provider's eligible patients screened for lung cancer, use of the tool, patient knowledge and satisfaction from patient surveys).
  Academic Detailing: All sites will be offered an academic detailing approach to implementation of Lung Decision Precsion. A trained detailer will travel to all sites who agree to a visit. The detailer will meet with individual primary care providers whenever possible, and groups of providers as necessary. He will present evidence for a risk-based approach to screening and how to use the tool with patients to make tailored screening recommendations.
Arm/Group | Standard Implementation | Intensive Implementation
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Formative Evaluation to Determine the Factors Most Important for Successful Implementation of Decision Precision Tool
Description: Qualitative analysts will conduct telephone interviews with providers at each site who identify themselves as participating in shared decision making process with patients regarding lung cancer screening. Reporting for this report is number of interviews completed of number interviews requested.
Time Frame: At least one year post-implementation of Lung Decision Precision web-site
Population: Of sites randomized to each Arm, the number of providers involved in lung cancer screening who were completed an interview about DecisionPrecision and the risk-based approach of the number of providers who were asked to complete an interview.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Implementation | Intensive Implementation
Number analyzed (Participants) | 48 | 40
Participants | 25 | 13

ADVERSE EVENTS:
Time Frame: Adverse event data were not systematically collected. The intervention involved staff training and no contact with Veteran participants.
Description: Adverse event data were not systematically collected. The intervention involved staff training and no contact with Veteran participants. We maintained a log of any participant complaints for the duration of the project. There were a total of 3, but we do not know which group the participants were in. The group was determined by which facility the Veteran received care from. Had there been a breach of data, we would have considered this an adverse event.
Arm/Group | Standard Implementation | Intensive Implementation
All-Cause Mortality (participants affected / at risk) | 482/5275 | 855/11758
Serious Adverse Events (participants affected / at risk) | 0/5275 | 0/11758
Other Adverse Events (participants affected / at risk) | 0/5275 | 0/11758

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT02765412/Prot_SAP_000.pdf